CLINICAL TRIAL: NCT02044536
Title: Retrospective Study of Current Practice Pattern and Effect of Training in Upper Endoscopic Biopsy
Brief Title: Current Practice Pattern and Effect of Training in Upper Endoscopic Biopsy
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, Department of Gastroenterology, Doctor, Chuncheon Sacred Heart Hospital
Other Study IDs: BCS-2
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Neoplasm
Keywords: biopsy; endoscopy; neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Faculty doctors: Experienced endoscopists (> 6000 cases). no intervention
  Interventions: Other: No intervention
- Trainees: Doctors on fellowship who are inexperienced endoscopists (< 4 months of endoscopy training) no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — retrospective data review

SUMMARY:
The optimal number of biopsy and the detection rate of neoplastic lesions are not established. The aim of this study is to assess the current practice pattern and effect of training in upper endoscopic biopsy.

DETAILED DESCRIPTION:
The endoscopic examination is indicated in the diagnosis of variety of gastrointestinal diseases and screening for the neoplastic lesions. Especially, in Korea where the stomach cancer prevalent area, high-quality endoscopic examination is required not to overlook pathologic lesions. Endoscopic biopsy is the gold standard for the confirmation of endoscopic diagnosis. It is usually decided based on the abnormal morphology of the lesions or color change of the mucosa. Diagnostic accuracy is known to be improved by training or using optical techniques or chromoendoscopy. With the development of endoscopic imaging technologies such as narrow band imaging (NBI), confocal imaging or magnifying techniques, the diagnostic accuracy can be enhanced. However, inspection with conventional white light endoscopy is still the most prevalent and basic form of screening or surveillance endoscopy. Thus, detecting lesions by meticulous inspection and accurate approach by targeted biopsy are important for the diagnosis of pathologic lesions. However, the optimal number of biopsy and the detection rate of neoplastic lesions are not established. This study aimed at evaluating the current practice pattern and effect of training in conventional upper endoscopic biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic EGD including screening endoscopy for health check-up or endoscopic examinations for the symptomatic patients to make a diagnosis.

Exclusion Criteria:

* Specimens from therapeutic procedures, such as endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From May to July 2013, all the biopsy specimens from diagnostic esophagogastroduodenoscopy will be collected and analyzed in a single teaching hospital of Korea.
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Concordance rate of endoscopic diagnosis and histologic diagnosis | During 3 months (retrospective endoscopy data review)
  In the evaluation of concordance rate and discrepancy rate, endoscopic diagnosis in the procedure report and histologic diagnosis in the pathology report will be compared.

SECONDARY OUTCOMES:
Neoplastic lesion detection rate | During 3 months (retrospetive endoscopy data review)
  Neoplasm detection rates of diagnostic upper endoscopic biopsy between trainees and faculty doctors will be compared statistically.

OTHER OUTCOMES:
Distribution of the biopsied lesion | During 3 months (retrospective endoscopy data review)
  The distribution of the histologic and endoscopic diagnosis for total biopsied lesion will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, Principal Investigator — Department of Internal Medicine, Hallym University College of Medicine, Korea
Locations (1):
- Department of Internal Medicine, Chuncheon Sacred Heart Hospital, Hallym University College of Medicine, Chuncheon, Gangwon-do, South Korea